CLINICAL TRIAL: NCT06821516
Title: Comparison of Analgesic Effectiveness Between Pericapsular Nerve Group (PENG) Block and Lumbar Erector Spinae Plane Block in Patients Undergoing Total Hip Arthroplasty With Spinal Anesthesia: a Randomized Controlled Trial
Brief Title: Comparison of Pain Relief Methods for Hip Surgery: A Study on Two Different Nerve Block Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Muzaffer GENCER, Associate Professor Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSH-ANES-BS-01
Record Dates: First submitted 2025-01-28; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Opioid Consumption, Postoperative; Pain, Postoperative; Nerve Block; PENG Block; Lumbar Erector Spinae Plane Block; Hip Replacement, Total; Postoperative Analgesia
Keywords: Pericapsular Nerve Group (PENG) Block; Lumbar Erector Spinae Plane Block; Total Hip Arthroplasty; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Patients who are admitted to the orthopedic and traumatology clinic and are scheduled for total hip arthroplasty surgery will be informed and monitored prior to the operation under spinal anesthesia. Preoperatively, either Pericapsular Nerve Group Block (PENG) (Group P) or Lumbar Erector Spina Plane Block (Group E) will be applied. Randomization will be performed using a computer-based method (http://www.randomizer.org) with a 1:1 allocation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants undergoing total hip arthroplasty with preoperative PENG block (Active Comparator)
  Interventions: Procedure: Evaluation of the postoperative analgesic effectiveness of PENG block in participants undergoing total hip arthroplasty under spinal anesthesia
- Participants undergoing total hip arthroplasty with preoperative Lumbar ESP block (Active Comparator)
  Interventions: Procedure: Evaluation of the postoperative analgesic effectiveness of lumbar erector spinae block in participants undergoing total hip arthroplasty under spinal anesthesia

INTERVENTIONS:
Procedure: Evaluation of the postoperative analgesic effectiveness of PENG block in participants undergoing total hip arthroplasty under spinal anesthesia — Evaluation of the postoperative analgesic effectiveness of PENG block in participants undergoing total hip arthroplasty under spinal anesthesia
  Arms: Participants undergoing total hip arthroplasty with preoperative PENG block
Procedure: Evaluation of the postoperative analgesic effectiveness of lumbar erector spinae block in participants undergoing total hip arthroplasty under spinal anesthesia — Evaluation of the postoperative analgesic effectiveness of lumbar erector spinae block in participants undergoing total hip arthroplasty under spinal anesthesia
  Arms: Participants undergoing total hip arthroplasty with preoperative Lumbar ESP block

SUMMARY:
This prospective randomized comparative study aims to compare the analgesic efficacy of pericapsular nerve group block (PENG) and lumbar erector spinae plane block (L-ESP) groups to relieve postoperative pain in participants over the age of 18 undergoing total hip arthroplasty under spinal anesthesia. The main question it aims to answer is:

To demonstrate whether PENG block or L-ESP block is more effective in postoperative analgesia in patients undergoing total hip arthroplasty surgery based on pain scores, opioid consumption, and patient satisfaction.

Total hip arthroplasties cause severe pain with movement in the postoperative period. After surgery, the movements of the participants are severely restricted, which increases the possibility of complications. In this study, the participants' pain status, VAS score, opioid consumption through patient-controlled analgesia, and patient satisfaction will be measured with a questionnaire for 24 hours at predetermined time points and then compared. Both types of blocks have pain-relieving effects. This study will only investigate which one is more effective in reducing pain, and there will be no deficiency in relieving the pain of the participants.

DETAILED DESCRIPTION:
Due to increasing life expectancy and the prevalence of obesity, hip arthroplasty surgeries have been steadily increasing, especially in the last twenty years, and these patients experience very serious postoperative pain. Postoperative pain control has a significant impact on earlier ambulation, initiation of physical therapy, better functional recovery, and patient satisfaction. At the same time, optimal pain management is of great importance in contributing to the reduction of the duration of hospital stay, the risk of adverse events such as deep vein thrombosis, and mortality.

Although peripheral nerve blocks have been shown to be effective as part of multimodal analgesia for successful postoperative pain management, the superiority of nerve blocks over each other in terms of analgesic efficacy is a subject of research.

This study was planned to show which of the Pericapsular Nerve Group (PENG) Block and Lumbar Erector Spina Plane Block to be applied to patients undergoing total hip arthroplasty is more effective in terms of postoperative effective analgesia duration, perioperative hemodynamic stability, reducing opioid dependence and postoperative delirium, reducing total opioid consumption, providing early mobilization and shortening the length of hospital stay.

Pericapsular nerve group (PENG) block is a promising regional analgesia procedure that protects the motor function of the hip joint by blocking the obturator nerve, femoral nerve and accessory obturator nerves by injecting local anesthetic between the superior pubic ramus and psoas muscle tendon. Erector spina plane block (ESPB) has been widely used at the thoracic vertebral level in 2016 with ultrasound-guided local anesthetic injection between the erector spinae muscle and the transverse process of the thoracic vertebra. In a single case study published in 2018, lumbar ESPB (L-ESPB) was used as postoperative analgesia after hip arthroplasty, and the local anesthetic injected from the fourth lumbar spine level (L4) spread to the cephalic and caudal directions and provided satisfactory hip analgesia.

Since both blocks are relatively newly defined blocks, there are limited studies in the literature and it is aimed to find an answer to the question of which of these two block types should be preferred by evaluating different parameters in providing postoperative analgesia in hip arthroplasty surgery.

Pericapsular Nerve Group Block (PENG) (Group P) or Lumbar Erector Spina Plane Block (Group E) will be applied preoperatively to patients hospitalized in the orthopedics and traumatology clinic who come to the operating room to undergo Total Hip Arthroplasty Surgery, after the necessary information is provided and monitoring is provided before being taken to the operation with spinal anesthesia. Randomization will be done 1:1 with a computer (using http://www.randomizer.org). Spinal anesthesia will be applied to patients who have preoperative block.

Patient-controlled analgesia (PCA) will be applied to all patients to evaluate opioid consumption at the end of the surgery. The patient's total opioid consumption will be recorded. Pain is a symptom known to be subjective and will be questioned with the Numeric Rating Scale (NRS), a standardized scale, in order to minimize differences between patients. At predetermined time points, Baseline 0, peroperative 15th minute, 1st hour, 2nd hour and postoperative 1st, 3rd, 6th, 12th, 24th hours, the patients' pain scores with the Numeric Rating Scale (NRS) (0-10; 0-3: mild pain, 4-6: moderate pain, 7-10: severe pain) will be questioned and noted. When the pain score is 4 and above, 20 mg tenoxicam will be administered as rescue analgesia and the total amount required will be recorded.

In both groups, patients' demographic data, ASA scores, surgery duration, hemodynamic parameters during the operation (systolic, diastolic blood pressure, mean arterial pressure, heart rate and SpO2 values), the time when the pain sensation started after the operation, the block termination process in the service follow-ups, the time when the additional analgesics was first needed, the dose administered, the numerical rating scale when the patient was asked to describe the pain intensity numerically, patient satisfaction scores (4: very satisfied, 3: satisfied, 2: less satisfied, 1: not satisfied), hospital stay, nausea-vomiting score and other complications related to the applied blocks will be recorded and followed for the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary willingness to participate in the study.
* Patients who will undergo Total Hip Arthroplasty surgery.
* Patients aged over 18 years.
* ASA score I-II-III.
* Patients who are fully oriented and can cooperate.

Exclusion Criteria:

* ASA score IV-V.
* Patients who refuse to participate in the study.
* Patients under 18 years of age.
* Presence of active infection in the area to be operated on.
* Chronic pain and continuous analgesic use.
* Patients with coagulation disorders.
* Patients who cannot cooperate with postoperative pain follow-up.
* Patients with allergies to local anesthetic agents.
* Presence of neuropathy or myopathy in the operated extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness on pain scores | at Baseline 0, perioperative 15th minute, 1st hour, 2nd hour, and postoperative 1st, 3rd, 6th, 12th, and 24th hours after preoperative peripheral nerve block
  Postoperative pain assessment is performed using the Numerical Rating Scale (NRS). Participants are asked about their rest pain at Baseline 0, perioperative 15th minute, 1st hour, 2nd hour, and postoperative 1st, 3rd, 6th, 12th, and 24th hours after applying a postoperative peripheral nerve block. With this method, participants rate their pain with a precise numerical value from 0 to 10. While zero(0) represents "no pain"; Ten (10) represents the opposite end of the pain continuum (e.g., "The most intense pain imaginable," "As intense pain as possible," "Maximum pain").

SECONDARY OUTCOMES:
Effect on total narcotic analgesic consumption | The total number of bolus doses administered by the intravenous PCA device at the end of 24 hours postoperatively
  After the surgery, patients will be given intravenous patient-controlled analgesia (PCA). "Tramadol" was preferred as the treatment method to be used for the PCA method. In preparation for PCA, 400 mg of tramadol is added to 100 cc of physiological saline. As PCA protocol, without basal infusion dose, 5 cc (20 mg) bolus dose, 20 minutes lockout period (maximum 3 bolus doses in 1 hour) are set. The total number of bolus doses administered by the participants on the PCA device at the end of 24 hours will be recorded and evaluated as the amount of additional opioid needed.
Time, frequency, and amount of rescue analgesia administration | first 24 hours postoperatively
  Pain scores (0-10; 0-3: mild pain, 4-6: moderate pain, 7-10: severe pain) will be questioned and noted with the Numerical Rating Scale (NRS). When the pain score is 4 and above, 20 mg tenoxicam will be administered as rescue analgesia and the total amount required will be recorded.
Time-dependent perioperative changes in preoperative blood pressure | Pre-block, post-block, perioperative 0th and 30th minutes, 1st and 2nd hours, and end of surgery
  Pre-block, post-block, perioperative 0th and 30th minutes, 1st and 2nd hours, and end of surgery blood pressure values will be noted.
Time of first mobilization | first 24 hours postoperatively
  Time of first mobilization will be noted.
Length of hospital stay | first 24 hours postoperatively
  Length of hospital stay will be noted.
Postoperative nausea and vomiting assessment | first 24 hours postoperatively
  Nausea-vomiting descriptive scale (0: none, 1: mild nausea, 2: nausea, 3: vomiting once, 4: vomiting more than once) will be noted and 0.1 mg/kg IV ondansetron will be administered for scores of 2 and above.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Çam Ve Sakura City Hospital, Istanbul, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Townsend D, Siddique N, Kimura A, Chein Y, Kamara E, Pope J, Weiser M, Nair S, Muse I. Lumbar Erector Spinae Plane Block for Total Hip Arthroplasty Comparing 24-Hour Opioid Requirements: A Randomized Controlled Study. Anesthesiol Res Pract. 2022 Oct 3;2022:9826638. doi: 10.1155/2022/9826638. eCollection 2022. PMID 36225251
- [Background] Medhat MM, Kamel AAF, Salem DAE, Alagamy SA, Fathi HM. The Analgesic Effects of Preemptive Ultrasound-Guided Pericapsular Nerve Group Block in Comparison with Erector Spinae Plane Block in Elderly Undergoing Hip Arthroplasty: A Randomized Controlled Trial. Anesth Pain Med. 2023 Sep 4;13(5):e138623. doi: 10.5812/aapm-138623. eCollection 2023 Oct. PMID 38028113
- [Background] Marrone F, Fusco P, Tulgar S, Paventi S, Tomei M, Fabbri F, Iacovazzi M, Pullano C. Combination of Pericapsular Nerve Group (PENG) and Sacral Erector Spinae Plane (S-ESP) Blocks for Hip Fracture Pain and Surgery: A Case Series. Cureus. 2024 Feb 7;16(2):e53815. doi: 10.7759/cureus.53815. eCollection 2024 Feb. PMID 38332999
- [Background] Pai P, Amor D, Lai YH, Echevarria GC. Use and Clinical Relevancy of Pericapsular Nerve Block (PENG) in Total Hip Arthroplasty: A Systematic Review and Meta-analysis. Clin J Pain. 2024 May 1;40(5):320-332. doi: 10.1097/AJP.0000000000001196. PMID 38268183
- [Background] Zheng J, Pan D, Zheng B, Ruan X. Preoperative pericapsular nerve group (PENG) block for total hip arthroplasty: a randomized, placebo-controlled trial. Reg Anesth Pain Med. 2022 Mar;47(3):155-160. doi: 10.1136/rapm-2021-103228. Epub 2021 Dec 6. PMID 34873023